CLINICAL TRIAL: NCT06857461
Title: Effect of the Uriclarity Program on the Perception of Insufficient Milk Supply in Postpartum Women From Three Hospitals in Piura-Peru Evaluated Through a Randomized Controlled Trial
Brief Title: Effect of the Uriclarity Program on Perceived Milk Supply in Postpartum Women in Piura-Peru
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Crianzamor (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 202500001
Record Dates: First submitted 2025-02-26; First posted 2025-03-04 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Perceived Insufficient Milk Supply
Keywords: Breastfeeding; Uriclarity Program; Perceived Insufficient Milk Supply; Lactation Support
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Uriclarity Program Group (Experimental): Participants in this arm will receive the Uriclarity Program, a structured lactation support intervention. The program includes a two-hour in-person workshop within the first 24-48 hours postpartum, covering breastfeeding education, self-monitoring using the Ashiyama Uriscale, and hands-on guidance. Right after discharge, participants will receive follow-up support via WhatsApp including educational videos.
  Interventions: Behavioral: Uriclarity Program
- Control Group (No Intervention): Participants in this arm will receive standard lactation counseling provided by hospital staff before discharge. This includes general breastfeeding guidance but does not involve hands-on training, structured self-monitoring tools, or follow-up support after hospital discharge.

INTERVENTIONS:
Behavioral: Uriclarity Program — The Uriclarity Program is a behavioral lactation support intervention designed to reduce the perception of insufficient milk supply (PIM) in postpartum women. The program consists of a two-hour hands-on training session delivered within the first 24-48 hours postpartum and a WhatsApp-based follow-up support system.
  During the in-person training, participants learn essential breastfeeding techniques, how to recognize normal lactation patterns, and how to use the Uriescala Ashiyama, a self-monitoring tool that evaluates neonatal urine color to assess milk transfer. Right after hospital discharge, participants receive virtual support including educational videos.
  This intervention differs from standard lactation counseling by integrating self-monitoring strategies, community-based digital support, and a non-technology-dependent educational approach, making it a scalable and sustainable strategy for breastfeeding promotion.
  Arms: Uriclarity Program Group

SUMMARY:
The goal of this clinical trial is to assess whether the Uriclarity Program is effective in reducing the perception of insufficient milk supply (PIM) in postpartum women. The study also aims to evaluate the feasibility of implementing this program as a lactation support strategy. The main research questions are:

Does the Uriclarity Program reduce the perception of insufficient milk supply among postpartum women? How does the program impact breastfeeding confidence and adherence to exclusive breastfeeding? Researchers will compare the Uriclarity Program to standard postpartum lactation counseling to determine its effectiveness.

Participants will:

Receive either the Uriclarity Program intervention or standard lactation counseling within 24-48 hours postpartum.

Be evaluated on days 1, 3, 7, and 14 postpartum using the PIM questionnaire to assess changes in perception.

Engage in follow-up via WhatsApp support groups (for the intervention group). This randomized controlled trial will provide evidence on whether the Uriclarity Program can effectively reduce maternal concerns about milk supply and support exclusive breastfeeding.

DETAILED DESCRIPTION:
This study is a randomized controlled trial (RCT) designed to evaluate the effect of the Uriclarity Program on the perception of insufficient milk supply (PIM) in postpartum women. The trial will be conducted in three hospitals in Piura, Peru between March and April 2025.

Study Rationale Perceived insufficient milk supply is a leading cause of early breastfeeding cessation, despite adequate milk production in most cases. The Uriclarity Program is a structured intervention aimed at enhancing maternal confidence in lactation by providing hands-on training and self-monitoring tools. This includes the Uriescala Ashiyama, a validated method that assesses neonatal urine color to help mothers monitor milk transfer.

Study Design Population: Postpartum women with term infants (37-41 weeks gestation) practicing exclusive breastfeeding.

Intervention Group: Receives the Uriclarity Program, consisting of a 2-hour hands-on training session, followed by WhatsApp-based follow-up support.

Control Group: Receives standard lactation counseling before hospital discharge.

Primary Outcome: Change in PIM scores at days 1, 3, 7, and 14 postpartum, assessed using a validated PIM questionnaire.

Sample Size: 40 participants per group (total 80 mothers), determined using a power analysis for proportion comparison.

Statistical Analysis Between-group comparison: Mann-Whitney U test for ordinal PIM scores. Longitudinal analysis: Mixed-effects ordinal logistic regression to evaluate PIM progression over time.

Confounder adjustment: Multivariable logistic regression, controlling for maternal age, parity, and education.

Significance This study seeks to provide high-quality evidence on a low-cost, scalable intervention that could reduce unnecessary formula supplementation and promote exclusive breastfeeding. If successful, the Uriclarity Program could be integrated into maternal care policies to support breastfeeding mothers.

ELIGIBILITY:
Inclusion Criteria:

* Postpartum women within 24-48 hours after delivery (vaginal or cesarean).
* Term neonates (37-41 weeks of gestation).
* Exclusive breastfeeding at enrollment.
* Maternal education level of at least primary school completed.
* Ability to use a smartphone with WhatsApp for follow-up support.

Exclusion Criteria:

* Maternal conditions that may affect breastfeeding, such as flat or inverted nipples, diabetes, hypertension, or morbid obesity.
* Maternal medication with effects on lactation.
* Cigarette smoking.
* Neonatal conditions impacting breastfeeding, including congenital heart defects, cleft lip/palate, or ankyloglossia.
* Use of infant formula, pacifiers, or bottles before enrollment.
* Diagnosed maternal or neonatal illness after study enrollment that may interfere with breastfeeding.
* Newborns who experienced hypoglycemia, weight loss equal to or greater than 7%, or any condition related to breastfeeding failure during their hospital stay.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2025-05-28 (Actual); Primary Completion 2025-08-24 (Actual); Study Completion 2025-08-24 (Actual)

PRIMARY OUTCOMES:
Reduction in Perceived Insufficient Milk Supply (PIM) Score | Baseline (Day 1), Day 3, Day 7, and Day 14 postpartum
  The Perceived Insufficient Milk Supply (PIM) Score will be assessed using a validated questionnaire at baseline (Day 1) and follow-ups on Days 3, 7, and 14 postpartum. A decrease in the PIM score indicates an improvement in maternal confidence regarding milk supply. The effect of the Uriclarity Program will be compared between the intervention and control groups.

CONTACTS AND LOCATIONS:
Overall Officials: Jackeline Ashiyama Vega, NP, Principal Investigator — Crianzamor
Locations (2):
- Peru (2):
  - Hospital de Chulucanas, Piura, Chulucanas
  - Crianzamor, Piura, Piura

IPD SHARING:
Plan to Share IPD: Yes
The following Individual Participant Data (IPD) will be shared:
  1. De-identified participant-level data for Perceived Insufficient Milk Supply (PIM) scores at baseline (Day 1), Day 3, Day 7, and Day 14 postpartum.
  2. Demographic variables (age, parity, education level).
  3. Intervention group assignment (Uriclarity Program vs. Control). Data will be available upon reasonable request for research purposes only, following ethical and regulatory guidelines.
Supporting Information: Study Protocol
Time Frame: IPD and supporting documents will be available starting 6 months after the primary results are published and will remain accessible for at least 1 year.
Access Criteria: De-identified Individual Participant Data (IPD) and supporting documents will be accessible to qualified researchers affiliated with academic institutions, research organizations, or healthcare agencies.
  Researchers must submit a formal request, including a study proposal and ethical approval, to the principal investigator. Upon approval, data will be shared via a secured repository or institutional data-sharing agreement.
  Data will be available for secondary analysis, systematic reviews, and meta-analyses, but not for commercial use or participant re-identification.

REFERENCES:
- [Background] Rodrigo R, Rodrigo A, Liyanage N, Hatahagoda W, Hewavitharana U. Maternal Perception of Adequacy of Mother's Milk Among Mothers Giving Birth at a Teaching Hospital in Sri Lanka. J Hum Lact. 2019 Feb;35(1):171-180. doi: 10.1177/0890334418773304. Epub 2018 May 22. PMID 29787682
- [Background] Peacock-Chambers E, Dicks K, Sarathy L, Brown AA, Boynton-Jarrett R. Perceived Maternal Behavioral Control, Infant Behavior, and Milk Supply: A Qualitative Study. J Dev Behav Pediatr. 2017 Jul/Aug;38(6):401-408. doi: 10.1097/DBP.0000000000000455. PMID 28570412
- [Background] Gatti L. Maternal perceptions of insufficient milk supply in breastfeeding. J Nurs Scholarsh. 2008;40(4):355-63. doi: 10.1111/j.1547-5069.2008.00234.x. PMID 19094151
- [Background] Huang Y, Liu Y, Yu XY, Zeng TY. The rates and factors of perceived insufficient milk supply: A systematic review. Matern Child Nutr. 2022 Jan;18(1):e13255. doi: 10.1111/mcn.13255. Epub 2021 Aug 12. PMID 34382733
- [Background] Victora CG, Bahl R, Barros AJ, Franca GV, Horton S, Krasevec J, Murch S, Sankar MJ, Walker N, Rollins NC; Lancet Breastfeeding Series Group. Breastfeeding in the 21st century: epidemiology, mechanisms, and lifelong effect. Lancet. 2016 Jan 30;387(10017):475-90. doi: 10.1016/S0140-6736(15)01024-7. PMID 26869575